CLINICAL TRIAL: NCT03694483
Title: Quantification and Purification of Circulating Prostasomes as Diagnostic Tool for Prostate Cancer Detection
Brief Title: Prostasomes as Diagnostic Tool for Prostate Cancer Detection
Status: Suspended | Type: Observational
Why Stopped: Staffing changes, pending funding renewal
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Uppsala University, Sweden (Department of Immunology, Genetics and Pathology) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro2018-0517
Record Dates: First submitted 2018-09-25; First posted 2018-10-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: prostasomes,; prostate cancer,; biomarkers
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient population: Male individuals with elevated PSA and a positive MRI-driven biopsy AND male individuals with diagnosed prostate cancer (but prior to any treatment)
  Interventions: Diagnostic Test: Genetic analysis for the detection of prostasomes
- Control Population: Male individuals with elevated PSA and a negative MRI-driven biopsy
  Interventions: Diagnostic Test: Genetic analysis for the detection of prostasomes

INTERVENTIONS:
Diagnostic Test: Genetic analysis for the detection of prostasomes — Whole blood will be collected and processed within 2 hours. Samples will be brought to Hackensack University Medical Center and will be centrifuged.
  The plasma samples will be tested for presence of prostasomes using the ExoPLA (Exosome in situ Proximity Ligation Assay) assay and the prostasomes will be purified for further miRNA sequencing.

SUMMARY:
Prostate cancer is the most frequently diagnosed cancer among men over 50 years old in Western societies, with an incidence that is steadily increasing in most countries. The current, most commonly used biomarker for prostate cancer is prostate specific antigen (PSA), which has well known limitations in accuracy and requires additional testing. However, prostate cancer cells secrete exosomes, also known as prostasomes, which are only detectable in the blood of prostate cancer patients. The presence of prostasomes in the blood is in itself a prostate cancer diagnosis. However, the assay that has been designed for the purification of prostasomes requires additional testing for evaluating its robustness and usefulness in the clinical setting. Additionally, the evaluation of the cargo of the purified prostasomes may provide more information on the nature of the prostate cancer, which may help develop a molecular assay for a prostate cancer liquid biopsy rather than a tissue biopsy. Therefore, the purpose of this study is two-fold: a validation phase where the purification of prostasomes will be tested on plasma collected from prostate cancer patients and a molecular testing phase where the contents of the purified prostasomes will be evaluated on their ability to determine the grade of the prostate tumors.

We will collaborate with Dr. Masood Kamali-Moghaddam at the Uppsala University (Department of Immunology, Genetics and Pathology) for molecular assay processing.

ELIGIBILITY:
Inclusion Criteria:

* Male
* With elevated PSA or patients with diagnosed prostate cancer
* 18 years and older
* Willingness to participate in the study and compliance with protocol requirements
* Have not received any type of treatment for prostate cancer

Exclusion Criteria:

* Patients with confirmed or suspected prostate cancer that have already received any type of treatment
* Patients with another primary cancer within the past five years of prostate cancer diagnosis. However, superficial skin cancers such as basal cell or squamous cell cancers would not exclude a patient.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All male patients with elevated PSA and suspected for prostate cancer or patients with diagnosed prostate cancer but prior to treatment will be invited to participate. Depending on the results from the diagnostic MRI-guided biopsy, participants will be assigned to either the control cohort (if biopsy is negative) or the patient cohort (if biopsy is positive).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity of the prostasome purification methodology | through study completion - up to 24 months
  true positive rate of the prostasomes purification methodology using the prostasome detection results for each of the patient specimens (cases and controls)
specificity of the prostasome purification methodology | through study completion - up to 24 months
  true negative rate of the prostasomes purification methodology using the prostasome detection results for each of the patient specimens (cases and controls)

SECONDARY OUTCOMES:
Quantification of the miRNA expression profiles of the purified protostomes both before and after treatment (in patients cohort only) | through study completion - up to 24 months
  identify the top 20 most frequently expressed miRNA markers and their level of expression in each of the case patient specimens
Time to disease progression(in patient cohort only) | Up to 24 months
Time to disease relapse (in patient cohort only) | Up to 24 months
Overall survival (in patient cohort only) | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Gomella LG, Johannes J, Trabulsi EJ. Current prostate cancer treatments: Effect on quality of life. Urology. 2009;73(5, Suppl): S28-S35. 2. Network, N.C.C. NCCN Clinical Practice Guidelines in Oncology: Prostate Cancer, Version 2.2017. [cited 2017 May 31];2017 Available from: https://www.nccn.org/professionals/physician_gls/pdf/prostate.pdf. 3. Pienta KJ. Critical appraisal of prostate-specific antigen in prostate cancer screening: 20 years later. Urology. 2009;73(5, Suppl):S11-S20. 4. Stamey TA, et al. Prostate-specific antigen as a serum marker for adenocarcinoma of the prostate. N Engl J Med. 1987;317:909-916. 5. Catalona WJ. Management of cancer of the prostate. N Engl J Med. 1994;331:996-1004. 6. Harvey P, et al. A systematic review of the diagnostic accuracy of prostate specific antigen. BMC Urol. 2009;9:14. 7. Cramer SD, et al. Association between genetic polymorphisms in the prostate-specific antigen gene promoter and serum prostate-specific antigen levels. J Natl Cancer Inst. 2003;95:1044-1053.
- [Background] 8. Inal JM, Kosgodage U, Azam S, Stratton D, Antwi-Baffour S, Lange S. Blood/plasma secretome and microvesicles. Biochim Biophys Acta. 2013;1834(11):2317-25. 9. Ronquist G, Brody I, Gottfries A, Stegmayr B. An Mg2+ and Ca2+-stimulated adenosine triphosphatase in human prostatic fluid-part II. Andrologia. 1978;10:427-433. 10. Ronquist G, Brody I, Gottfries A, Stegmayr B. An Mg2+ and Ca2+-stimulated adenosine triphosphatase in human prostatic fluid: Part I. Andrologia. 1978;10:261-272. 11. Ronquist G, Hedström M. Restoration of detergent-inactivated adenosine triphosphatase activity of human prostatic fluid with concanavalin A. Biochim Biophys Acta. 1977;483:483-486. 12. Minciacchi VR, Zijlstra A, Rubin MA, Di Vizio D. Extracellular vesicles for liquid biopsy in prostate cancer: where are we and where are we headed? Prostate Cancer Prostatic Dis. 2017;20(3):251-258. 13. Poliakov A, Spilman M, Dokland T, Amling CL, Mobley JA. Structural heterogeneity and protein composition of exosome-like vesicles (prostasomes) in human semen. Prostate. 2009;69:159-167. 14. Utleg AG, et al. Proteomic analysis of human prostasomes. Prostate. 2003;56:150-161. 15. Carlsson L, et al. Characteristics of human prostasomes isolated from three different sources. Prostate. 2003;54:322-330.
- [Background] 16. Carlsson L, Ronquist G, Eliasson R, Egberg N, Larsson A. Flow cytometric technique for determination of prostasomal quantity, size and expression of CD10, CD13, CD26 and CD59 in human seminal plasma. Int J Androl. 2006;29:331-338. 17. Fernández JA, Heeb MJ, Radtke KP, Griffin JH. Potent blood coagulant activity of human semen due to prostasome-bound tissue factor. Biol Reprod. 1997;56:757-763. 18. Fabiani R, Johansson L, Lundkvist O, Ronquist G. Enhanced recruitment of motile spermatozoa by prostasome inclusion in swim-up medium. Hum Reprod. 1994;9:1485-1489. 19. Carlsson L, Påhlson C, Bergquist M, Ronquist G, Stridsberg M. Antibacterial activity of human prostasomes. Prostate. 2000;44:279-286. 20. Rooney IA, et al. Physiologic relevance of the membrane attack complex inhibitory protein CD59 in human seminal plasma: CD59 is present on extracellular organelles (prostasomes), binds cell membranes, and inhibits complement-mediated lysis. J Exp Med. 1993;177:1409-1420. 21. Saez F, Motta C, Boucher D, Grizard G. Antioxidant capacity of prostasomes in human semen. Mol Hum Reprod. 1998;4:667-672. 22. Skibinski G, Kelly RW, Harkiss D, James K. Immunosuppression by human seminal plasma-extracellular organelles (prostasomes) modulate activity of phagocytic cells. Am J Reprod Immunol. 1992;28:97-103.
- [Background] 23. Floryk D, Tollaksen SL, Giometti CS, Huberman E. Differentiation of human prostate cancer PC-3 cells induced by inhibitors of inosine 5'-monophosphate dehydrogenase. Cancer Res. 2004;64:9049-9056. 24. Nilsson BO, Egevad L, Jin M, Ronquist G, Busch C. Distribution of prostasomes in neoplastic epithelial prostate cells. Prostate. 1999;39:36-40. 25. Sahlén G, et al. Prostasomes are secreted from poorly differentiated cells of prostate cancer metastases. Prostate. 2004;61:291-297. 26. Fredriksson S, et al. Protein detection using proximity-dependent DNA ligation assays. Nat Biotechnol. 2002;20:473-477. 27. Tavoosidana G, Ronquist G, Darmanis S, Yan J, Carlsson L, Wu D, Conze T, Ek P, Semjonow A, Eltze E, Larsson A, Landegren UD, Kamali-Moghaddam M. Multiple recognition assay reveals prostasomes as promising plasma biomarkers for prostate cancer. Proc Natl Acad Sci U S A. 2011 May 24;108(21):8809-14. 28. Löf L, Ebai T, Dubois L, Wik L, Ronquist KG, Nolander O, Lundin E, Söderberg O, Landegren U, Kamali-Moghaddam M. Detecting individual extracellular vesicles using a multicolor in situ proximity ligation assay with flow cytometric readout. Sci Rep. 2016; 6:34358. 29. Loudig O, Wang T, Ye K, Lin J, Wang Y, Ramnauth A, Liu C, Stark A, Chitale D, Greenlee R, Multerer D, Honda S, Daida Y, Spencer Feigelson H, Glass A, Couch FJ, Rohan T, Ben-Dov IZ. Evaluation and Adaptation of a Laboratory-Based cDNA Library Preparation Protocol for Retrospective Sequencing of Archived MicroRNAs from up to 35-Year-Old Clinical FFPE Specimens. Int J Mol Sci. 2017; 18(3). pii: E627. 30. Loudig O, Liu C, Rohan T, and Ben-Dov IZ. Retrospective MicroRNA Sequencing: Complementary DNA Library Preparation Protocol Using Formalin-fixed Paraffin-embedded RNA Specimens. Journal of Visualized Experiments, 2018.